CLINICAL TRIAL: NCT02407743
Title: Finding Good TEMporal PostOperative Pain Signatures (TEMPOS)
Brief Title: TEMporal PostOperative Pain Signatures
Acronym: TEMPOS
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201500153 -N; 1R01GM114290-01 (NIH); OCR18877 (Other: OnCore)
Record Dates: First submitted 2015-03-09; First posted 2015-04-03 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
Keywords: postoperative pain; surgery; pain resolution; pain intensity; persistent postsurgical pain; pain-related genes; analgesic
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Genetic Markers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical patients' clinical progression: Patients undergoing non-ambulatory surgery will be asked questions and complete surveys in an effort to characterize postoperative pain experience profiles. A blood sample will be obtained for genetic markers exploring a variety of pain-related genes.
  Interventions: Behavioral: Surgical patients' clinical progression; Genetic: Genetic markers

INTERVENTIONS:
Behavioral: Surgical patients' clinical progression — Study the dynamic nature of pain
Genetic: Genetic markers — Research variants in genes related to pain sensitivity, analgesic sensitivity and opioid response

SUMMARY:
The purpose of this research study is to determine what causes pain after surgery to increase or decrease over time.

DETAILED DESCRIPTION:
Before surgery, study participants will be asked questions about age, gender, race/ethnicity, annual income, and education level. Study participants will also be questioned regarding prior pain experiences, their mood and how they think about pain. A small test tube of blood, a cheek swab or a saliva sample will be taken to see what genetic differences may influence individuals pain after surgery.

After surgery, study participants will be asked questions about their pain intensity while in the hospital. Additional information will be collected about the effects of pain medicine, and their recovery from surgery.

Following discharge from the hospital, study participants will be contacted monthly to confirm continued communication. Study participants will also be contacted six months after surgery, and asked to complete a final survey about their pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* anticipated length of hospital stay of 72 hours or greater
* expected post-operative survival greater than 6 months

Exclusion Criteria:

* < 18 years of age
* anticipated need for prolonged post-operative intubation (greater than 24 hours)
* urgent or emergent surgical procedure
* inability to understand or participate in questionnaires, surveys or data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Measure postoperative pain scores change with respect to time | up to 7 days
  Pain scores will be measured using previously established pain scale and Questionnaire

SECONDARY OUTCOMES:
Measure variables that contribute to postoperative pain scores | up to 6 months
  Variables: clinical, biological, psychological, and social factors
Measure timing patterns that may influence development of persistent postsurgical pain (PPP) | up to 6 months
  Different patterns of pain analgesia-pain cycles
Genetic testing | up to 1 day
  Specific single nucleotide polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Tighe, MD, Principal Investigator — Assistant Professor of Anesthesiology and Program Director, Perioperative Analytics Group Joint Assistant Professor of Orthopedics
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No